CLINICAL TRIAL: NCT02330822
Title: A Clinical and Experimental Study to Evaluate the Efficacy of Locally Applied Hyaluronic Acid in Bone Healing Following Dental Extraction
Brief Title: Role of Hyaluronic Acid in Bone Healing After Dental Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-OMFS-01-2015
Record Dates: First submitted 2015-01-01; First posted 2015-01-05 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Patients With Dental Extraction
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyaluronic Acid Group (Experimental): In this Group, Hyaluronic acid will be injected following extraction.
  Interventions: Drug: Hyaluronic Acid
- Traditional Extraction Group (No Intervention): In this group, traditional extraction procedures will be followed.

INTERVENTIONS:
Drug: Hyaluronic Acid — This material is going to be injected into the extraction socket in order to promote bone healing.
  Arms: Hyaluronic Acid Group

SUMMARY:
This is a randomized controlled trial with a split mouth design. Patients with an indication of lower dental extraction will be asked to join this research project at the Department of Oral and Maxillofacial Surgery at University of Damascus Dental School. Each patient whose case requires bilateral extraction, one side will serve as an experimental side, whereas the other side will serve as a control.

Participants should have symmetric teeth that need extraction in the lower jaw. Hyaluronic acid will be injected following extraction in one of the two sides with random allocation.

cone-beam computerized tomography (CBCT) images will be taken for each participant immediately post-extraction and at six months post-operatively.

DETAILED DESCRIPTION:
I- Clinical examination variables:

Buccolingual distance and distomesial distance will be measured for each participant at 2 assessment times: directly post-extraction and six months post-extraction.

II- Radiographic examination variables:

Linear measurements Vertical bone fill Bone mineral density

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* Symmetric teeth requiring extraction in the lower jaw
* Systematically healthy

Exclusion Criteria:

* Smokers
* Pregnancy (for female participants)
* Diabetic patients
* Patients with metabolic problems

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in bone mineral density (BMD) | (BMD) will be measured two times in this study: directly at the day of extraction and six months post-extraction.
  BMD is the amount of bone tissue in a certain volume of bone. This variable is going to be measured on CBCT images.
Vertical bone fill | This variable is going to be measured at 6 months post-extraction
  'Vertical bone fill' is the distance between the base of the extraction socket and cement-enamel junction directly after extraction and minus the distance between base of the extraction socket and cement-enamel junction six months post-extraction.
  This variable is going to be measured on CBCT images.

SECONDARY OUTCOMES:
Buccolingual distance | at six months post-extraction
  Buccolingual distance is the distance between buccal wall and lingual wall of the extraction socket. This variable is going to be measured clinically.
Mesiodistal distance | at six months post-extraction
  Mesiodistal distance is the distance between mesial wall and distal wall of the extraction socket. This variable is going to be measured clinically.

CONTACTS AND LOCATIONS:
Overall Officials: Sireen Abu Atta, DDS MSc, Principal Investigator — PhD student, Department of Oral and Maxillofacial Surgery, University of Damascus Dental School; Mazen Zenati, DDS MSc PhD, Study Director — Professor of Oral and Maxillofacial Surgery, University of Damsacus Dental School
Locations (1):
- Department of Oral and Maxillofacial Surgery, University of Damascus Dental School, Damascus, Damscus, Syria

REFERENCES:
- [Background] Baldini A, Zaffe D, Nicolini G. Bone-defects healing by high-molecular hyaluronic acid: preliminary results. Ann Stomatol (Roma). 2010 Jan;1(1):2-7. Epub 2010 Jun 29. PMID 22238698
- [Background] Cardaropoli G, Araujo M, Hayacibara R, Sukekava F, Lindhe J. Healing of extraction sockets and surgically produced - augmented and non-augmented - defects in the alveolar ridge. An experimental study in the dog. J Clin Periodontol. 2005 May;32(5):435-40. doi: 10.1111/j.1600-051X.2005.00692.x. PMID 15842256
- [Background] de Brito Bezerra B, Mendes Brazao MA, de Campos ML, Casati MZ, Sallum EA, Sallum AW. Association of hyaluronic acid with a collagen scaffold may improve bone healing in critical-size bone defects. Clin Oral Implants Res. 2012 Aug;23(8):938-42. doi: 10.1111/j.1600-0501.2011.02234.x. Epub 2011 Jun 21. PMID 21689163